CLINICAL TRIAL: NCT02308137
Title: Open-label, Single-center, Single-arm Futility Trial Evaluating Oral Domperidone 10mg QID for Reducing Progression of Disability in Patients With Secondary Progressive Multiple Sclerosis (SPMS)
Brief Title: Domperidone in Secondary Progressive Multiple Sclerosis (SPMS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Alberta Innovates Health Solutions (Other)
Responsible Party: Principal Investigator, Dr. Marcus Werner Koch, Neurologist, Assistant Professor, University of Calgary
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Domperidone_MS01
Record Dates: First submitted 2014-12-02; First posted 2014-12-04 (Estimated); Last update posted 2020-02-24 (Actual); Status verified 2020-02

CONDITIONS: Multiple Sclerosis, Secondary Progressive
MeSH Terms: conditions — Multiple Sclerosis, Chronic Progressive | interventions — Domperidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Domperidone (Experimental): Treatment: Oral domperidone four times daily Target dose: 40mg per day Duration: 1 year
  Interventions: Drug: Domperidone

INTERVENTIONS:
Drug: Domperidone — Simon-2-stage design for domperidone futility
  Other Names: domperidone maleate

SUMMARY:
The purpose of this clinical trial is to determine if Domperidone in a dose of 40 mg daily can prevent worsening of walking ability in people secondary progressive MS. The number of participants in this study will be 62. A maximum of 75 people with secondary progressive MS will be included. Each patient will be followed for 12 months from inclusion. Domperidone is a medication which has been shown to increase levels of the hormone prolactin. The best understood function of prolactin is the stimulation of milk production in women after delivery. However, the increase in prolactin levels seen in patients treated with standard doses of Domperidone (in doses of up to 80mg per day) usually does not lead to clinical symptoms. Prolactin has been shown to improve myelin repair in mice. Domperidone therefore may also improve myelin repair in people with MS. Domperidone is currently approved in Canada to treat slow moving bowels and nausea, for instance in patients with Parkinson's Disease or Diabetes Mellitus, where too slowly moving bowels can cause constipation. Domperidone is available as a tablet that is usually taken four times per day. Doses up to 80mg per day may be used but we estimate that a dose of only 40mg daily will be needed to stimulate myelin repair. Domperidone is usually well tolerated.

DETAILED DESCRIPTION:
Primary objective

To demonstrate non-futility of domperidone for reducing progression of disability, as measured with the timed 25 foot walk (T25FW), in secondary progressive Multiple Sclerosis (SPMS).

Secondary objectives

* To assess the safety of domperidone in the study population for the duration of the study.
* To assess the effect of domperidone on hand dexterity as measured with the 9HPT
* To assess the effect of domperidone on cognition, as measured with the SDMT
* To assess the effect of domperidone on health related quality of life, as measured with the MSQOL-54
* To assess the effect of domperidone on fatigue, as measured with the MFIS
* To establish the Simon-2-stage model as a study model in MS research. The application of this methodology to studies in progressive MS will have important consequences for the design and conduct of clinical and translational research in progressive MS, in particular for phase II trials in progressive MS

ELIGIBILITY:
Inclusion Criteria:

* written informed consent obtained
* with Multiple Sclerosis, and with secondary progressive disease course
* screening Expanded Disability Status Scale (EDSS) score between 4.0 and 6.5 inclusive
* screening timed 25 foot walk (average of two trials) lof 9 seconds or more

Exclusion Criteria:

* Long QT interval, defined as corrected QT interval of more than 470 msec in men and more than 450 msec in women on baseline ECG
* Patients with known long-QT syndrome
* Patients with known ventricular arrhythmia
* Patients with a known electrolyte disturbance
* Patients undergoing treatment with drugs that increase the QTc interval
* Patients undergoing treatment with drugs that inhibit CYP3A4, in particular: Ketoconazole, Fluconazole, Erythromycin, Clarithromycin, Ritonavir
* Patients with a history of breast cancer or carcinoma in situ
* Patients with known renal insufficiency
* Patients with known allergy or other intolerability to domperidone
* Patients currently using Fampridine or 4-aminopyridine
* Patients planning to start Fampridine or 4-aminopyridine during the study period
* Patients planning to start Baclofen or Tizanidine during the duration of the study
* Patients planning to increase or decrease their dose of Baclofen or Tizanidine during the study period
* Patients planning to receive treatment with Botulinum toxin in the leg muscles during the duration of the study
* Patients with a significiant hepatic impairment
* Patients with a prolactinoma
* Patients in whom gastrointestinal stimulation could be dangerous
* Patients using MAO inhibitors
* Patients with a history of breast cancer
* Pregnant or breast-feeding women

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2020-01-03 (Actual); Study Completion 2020-01-03 (Actual)

PRIMARY OUTCOMES:
Timed 25-Foot Walk (T25W) | up to 12 months
  quantitative ambulation performance test

SECONDARY OUTCOMES:
9-Hole Peg Test | administered at baseline, one month, 6 months, and 12 months
  brief, standardized, quantitative test of upper extremity
Symbol Digit Modalities Test | administered at baseline, one month, 6 months, and 12 months
  measures cognitive processing speed and working memory
Functional Systems and Expanded Disability Status Scale (EDSS) | administered at baseline, one month, 6 months, and 12 months
  EDSS is the standard measure of neurologic impairment that is used to describe disability in MS. The neurological assessment comprises seven functional systems.
Modified Fatigue Impact Scale (MFIS) | administered at baseline, one month, 6 months, and 12 months
  structured, self-report questionnaire with 21 itmes concerning how fatigue impacts patient's life
Multiple Sclerosis Quality of Life Scale 54 item version | administered at baseline, one month, 6 months, and 12 months
  54-item multidimensional health-related quality of life measure that combines both generic and MS-specific items

CONTACTS AND LOCATIONS:
Overall Officials: Marcus W Koch, MD, PhD, Principal Investigator — University of Calgary
Locations (1):
- Calgary MS Clinic at Foothills Medical Centre, Calgary, Alberta, Canada

REFERENCES:
- [Background] Noseworthy JH, Lucchinetti C, Rodriguez M, Weinshenker BG. Multiple sclerosis. N Engl J Med. 2000 Sep 28;343(13):938-52. doi: 10.1056/NEJM200009283431307. No abstract available. PMID 11006371
- [Background] Nylander A, Hafler DA. Multiple sclerosis. J Clin Invest. 2012 Apr;122(4):1180-8. doi: 10.1172/JCI58649. Epub 2012 Apr 2. PMID 22466660
- [Background] Weinshenker BG, Bass B, Rice GP, Noseworthy J, Carriere W, Baskerville J, Ebers GC. The natural history of multiple sclerosis: a geographically based study. 2. Predictive value of the early clinical course. Brain. 1989 Dec;112 ( Pt 6):1419-28. doi: 10.1093/brain/112.6.1419. PMID 2597989
- [Background] Lassmann H, van Horssen J, Mahad D. Progressive multiple sclerosis: pathology and pathogenesis. Nat Rev Neurol. 2012 Nov 5;8(11):647-56. doi: 10.1038/nrneurol.2012.168. Epub 2012 Sep 25. PMID 23007702
- [Background] Rovaris M, Confavreux C, Furlan R, Kappos L, Comi G, Filippi M. Secondary progressive multiple sclerosis: current knowledge and future challenges. Lancet Neurol. 2006 Apr;5(4):343-54. doi: 10.1016/S1474-4422(06)70410-0. PMID 16545751
- [Background] Patrikios P, Stadelmann C, Kutzelnigg A, Rauschka H, Schmidbauer M, Laursen H, Sorensen PS, Bruck W, Lucchinetti C, Lassmann H. Remyelination is extensive in a subset of multiple sclerosis patients. Brain. 2006 Dec;129(Pt 12):3165-72. doi: 10.1093/brain/awl217. Epub 2006 Aug 18. PMID 16921173
- [Background] Franklin RJ, ffrench-Constant C, Edgar JM, Smith KJ. Neuroprotection and repair in multiple sclerosis. Nat Rev Neurol. 2012 Nov 5;8(11):624-34. doi: 10.1038/nrneurol.2012.200. Epub 2012 Oct 2. PMID 23026979
- [Background] Tselis A, Khan OA, Lisak RP. Approaches to neuroprotective strategies in multiple sclerosis. Expert Opin Pharmacother. 2010 Dec;11(17):2869-78. doi: 10.1517/14656566.2010.508070. Epub 2010 Aug 5. PMID 20687779
- [Background] Zhornitsky S, Yong VW, Weiss S, Metz LM. Prolactin in multiple sclerosis. Mult Scler. 2013 Jan;19(1):15-23. doi: 10.1177/1352458512458555. Epub 2012 Aug 29. PMID 22933621
- [Background] Rudick R, Antel J, Confavreux C, Cutter G, Ellison G, Fischer J, Lublin F, Miller A, Petkau J, Rao S, Reingold S, Syndulko K, Thompson A, Wallenberg J, Weinshenker B, Willoughby E. Recommendations from the National Multiple Sclerosis Society Clinical Outcomes Assessment Task Force. Ann Neurol. 1997 Sep;42(3):379-82. doi: 10.1002/ana.410420318. PMID 9307263
- [Derived] Koch MW, Sage K, Kaur S, Kim J, Cerchiaro G, Yong VW, Cutter GR, Metz LM. Repurposing Domperidone in Secondary Progressive Multiple Sclerosis: A Simon 2-Stage Phase 2 Futility Trial. Neurology. 2021 May 4;96(18):e2313-e2322. doi: 10.1212/WNL.0000000000011863. Epub 2021 Mar 23. PMID 34038379